CLINICAL TRIAL: NCT01945970
Title: Randomized Double Blind Placebo Controlled Crossover Study to Assess the Effect of Black Tea on Flow-Mediated Dilation in Healthy, Non-tea Drinking Males
Brief Title: Effect of Black Tea on Vascular Function
Acronym: Heraclitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REF-BEV-1134
Record Dates: First submitted 2013-09-08; First posted 2013-09-19 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Vascular Function
Keywords: Vascular function; Flow mediated dilation; Tea
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Black tea extract (Experimental): Spray dried aqueous extract of a representative batch of black tea
  Interventions: Other: Black tea extract
- Positive control (Active Comparator): Spray dried aqueous extract of a batch of tea extract that has shown to improve FMD previously
  Interventions: Other: Positive control
- Placebo (Placebo Comparator): Food grade colouring, artificial tea flavour and an amount of caffeine matched to the caffeine in the Black tea extract
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Black tea extract — Black tea extract
  Arms: Black tea extract
Other: Positive control — Positive control
  Arms: Positive control
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Epidemiological studies indicate that regular consumption of three cups of black tea per day reduces the risk of stroke or myocardial infarction. In a number of previous nutrition intervention studies tea has been shown to improve vascular function as assessed by Flow Mediated Dilation (FMD).

DETAILED DESCRIPTION:
The current study tests a specific Black tea extract against a placebo in population that has previously show to be sensitive to the effect of black tea on Flow Mediated dilation. A tea extract that has previously been shown to improve FMD is included as the positive control.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy male volunteers with no history of cardiovascular disease
* Having body mass index (BMI) of between 18.0 and 30.0 kg/m2 (inclusive)
* Non-smokers (> 2 years)
* Non-tea drinkers (less or equal 1 cup/week)
* Limited alcohol intake (less or equal 21 units/week)
* Systolic blood pressure less or equal 160 mmHg and/or diastolic blood pressure less or equal 100 mmHg at screening
* Brachial artery can be imaged using ultrasound and at screening FMD value is within the expected range as judged by the PI
* Judged to be in good health on the basis of medical history, physical examination and routine laboratory tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, glucose, highly sensitive C-reactive protein).

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ghiadoni, MD, Principal Investigator — University of Pisa, Internal medicine
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Centro di Farmacologia Clinicaper la Sperimentazione dei Farmaci, Pisa, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 suitable subjects recruited from database
Pre-assignment Details: 30 subjects randomised
Groups:
- Black Tea - Positive Control - Placebo: Subjects treated in the order Black tea - wash out- Positive control - wash out - Placebo.
  Treatments each lasted one week and were separated by a one week washout.
- Black Tea - Placebo - Positive Control: Subjects treated in the order Black tea - wash out- Placebo control - wash out - Positive control.
  Treatments each lasted one week and were separated by a one week washout.
- Positive Control - Black Tea - Placebo: Subjects treated in the order Positive control - wash out - Black tea - wash out - Placebo.
  Treatments each lasted one week and were separated by a one week washout.
- Positive Control - Placebo - Black Tea: Subjects treated in the order Positive control - wash out - Placebo - wash out - Black tea.
  Treatments each lasted one week and were separated by a one week washout.
- Placebo- Positive Control - Black Tea: Subjects treated in the order Placebo - wash out - Positive control - wash out- Black tea.
  Treatments each lasted one week and were separated by a one week washout.
- Placebo - Black Tea - Positive Control: Subjects treated in the order Placebo - wash out - Black tea - wash out- Positive control.
  Treatments each lasted one week and were separated by a one week washout.
Period: Overall Study
Arm/Group | Black Tea - Positive Control - Placebo | Black Tea - Placebo - Positive Control | Positive Control - Black Tea - Placebo | Positive Control - Placebo - Black Tea | Placebo- Positive Control - Black Tea | Placebo - Black Tea - Positive Control
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross over study where all subjects recieved all treatments
Groups:
- Study Subjects: All six treatment orders combined
Arm/Group | Study Subjects
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 43 [30 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 30
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (2.4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 118 (12)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74 (8)

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation, Acute-upon-chronic, Black Tea
Description: Flow mediated dilation (FMD) measurement included the following steps:
  * 1 minute base scan to measure the baseline diameter of artery (Resting stage)
  * 5 minutes of forearm occlusion at 300±30 mmHg (cuff occlusion stage), just below the elbow 2-5 cm from antecubital crease)
  * 4 minutes FMD scan, which started immediately after release of occlusion (reactive hyperaemia stage)
  * When the artery had returned to baseline a second 1 minute scan was taken
  * 25 µg sublingual glyceryl trinitrate (GTN) was given to the subject
  * 5 minutes GTN scan to assess the endothelium-independent dilation FMD and response to GTN was calculated as maximal percent increase in diameter above baseline (mean value of measures obtained during 1 minute before cuff inflation).
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 8.
Population: Intention to treat
Measure: Least Squares Mean (Standard Deviation); unit: percentage of flow mediated dilation
Groups:
- Black Tea Beverage: Participant when they received Back Tea
- Placebo Beverage: Participants when the received Placebo
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, before consumption of test product | 4.24 (1.57) | 4.48 (1.92)
  Day 8, 2 hours post consumption of test product | 4.49 (1.88) | 4.87 (1.94)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis; Subject as random factor, baseline same period and mean baseline in both periods as covariates, and treatment, operator, and period as fixed effects; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.09 to 0.40] — Effect of black tea adjusted for placebo

2. Secondary Outcome: Flow Mediated Dilation, Acute, Black Tea
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 1
Population: Intention to treat
Measure: Least Squares Mean (Standard Deviation); unit: percentage of flow mediated dilation
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, before consumption of test product | 4.24 (1.57) | 4.48 (1.92)
  Day 1, 2 hours post consumption of test product | 4.50 (1.89) | 4.13 (1.91)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.24 to 1.28] — Effect of black tea adjusted for placebo

3. Secondary Outcome: Flow Mediated Dilation, Chronic, Black Tea
Description: as for outcome 1
Time Frame: From before consumption day 1 to before consumption day 8.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of flow mediated dilation
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, before consumption of test product | 4.24 (1.57) | 4.48 (1.92)
  Day 8, before consumption of test product | 3.90 (1.67) | 4.84 (1.96)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.59 to -0.19] — Effect of black tea adjusted for placebo

4. Secondary Outcome: Flow Mediated Dilation, Acute-upon-chronic, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 8
Population: Intention to treat
Measure: Least Squares Mean (Standard Deviation); unit: percentage of flow mediated dilation
Groups:
- Positive Control Beverage: Participant when they received the positive control
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, before consumption of test product | 3.28 (1.67) | 4.48 (1.92)
  Day 8, 2 hours post consumption of test product | 4.21 (1.54) | 4.87 (1.94)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.22, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.49, 95% CI 2-sided [-1.30 to 0.31] — Effect of positive control adjusted for placebo

5. Secondary Outcome: Flow Mediated Dilation, Acute, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 1
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of flow mediated dilation
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, pre-consumption of test product | 3.28 (1.67) | 4.48 (1.92)
  Day 1, 2 hours post consumption of test product | 4.06 (1.78) | 4.13 (1.91)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.71, 95% CI 2-sided [-0.11 to 1.53] — Effect of positive control adjusted for placebo

6. Secondary Outcome: Flow Mediated Dilation, Chronic, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to before consumption day 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of flow mediated dilation
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of flow mediated dilation
  Day 1, pre-consumption of test product | 3.28 (1.67) | 4.48 (1.92)
  Day 8, pre-consumption of test product | 4.20 (1.65) | 4.84 (1.96)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.32, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.13 to 0.37] — Effect of positive control adjusted for placebo

7. Other Pre Specified Outcome: Systolic Blood Pressure, Black Tea
Description: Change in Systolic blood pressure
Time Frame: From before consumption on day 1 to before consumption on day 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Day 1, before consumption of test product | 111.7 (11.45) | 112.1 (10.75)
  Day 8, before consumption of test product | 113.7 (11.84) | 111.8 (10.41)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.14, Mixed Models Analysis; Subject as random factor and treatment and period as fixed effects; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-0.61 to 4.39] — Effect of black tea adjusted for placebo

8. Other Pre Specified Outcome: Diastolic Blood Pressure Black Tea
Description: Change in Diastolic blood pressure
Time Frame: From before consumption on day 1 to before consumption day 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Day 1, before consumption of test product | 72.23 (8.57) | 72.80 (8.07)
  Day 8, before consumption of test product | 71.77 (8.20) | 72.27 (8.38)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.69, Mixed Models Analysis; Subject as random factor and treatment and period as fixed effects; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-2.41 to 1.62] — Effect of black tea adjusted for placebo

9. Other Pre Specified Outcome: Systolic Blood Pressure, Positive Control
Description: Change in systolic blood pressure
Time Frame: From before consumption (baseline) day 1 to before consumption day 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Day 1, before consumption of test product | 112.9 (12.90) | 112.1 (10.75)
  Day 8, before consumption of test product | 112.3 (10.05) | 111.8 (10.41)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.72, Mixed Models Analysis; Subject as random factor and treatment and period as fixed effects; Median Difference (Final Values) = 0.44, 95% CI 2-sided [-2.06 to 2.95] — Effect of positive control adjusted for placebo

10. Other Pre Specified Outcome: Diastolic Blood Pressure, Positive Control
Description: Change in Diastolic Blood pressure
Time Frame: From before consumption on day 1 to before consumption day 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
mmHg
  Day 1, before consumption of test product | 72.00 (8.18) | 72.80 (8.07)
  Day 8, before consumption of test product | 72.98 (7.28) | 72.27 (8.38)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.39, Mixed Models Analysis; Subject as random factor and treatment and period as fixed effects; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-1.15 to 2.88] — Effect of positive control adjusted for placebo

11. Other Pre Specified Outcome: Endothelium Independent Dilation, Acute-upon-chronic, Black Tea
Description: FMD measurement included the following steps:
  * 1 minute base scan to measure the baseline diameter of artery (Resting stage)
  * 5 minutes of forearm occlusion at 300±30 mmHg (cuff occlusion stage), just below the elbow 2-5 cm from antecubital crease)
  * 4 minutes FMD scan, which started immediately after release of occlusion (reactive hyperaemia stage)
  * When the artery had returned to baseline a second 1 minute scan was taken
  * 25 µg sublingual glyceryl trinitrate (GTN) was given to the subject
  * 5 minutes GTN scan to assess the endothelium-independent dilation FMD and response to GTN was calculated as maximal percent increase in diameter above baseline (mean value of measures obtained during 1 minute before cuff inflation).
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 9.55 (3.81) | 9.67 (3.37)
  Day 8, 2 hours post consumption of test product | 9.02 (3.43) | 9.28 (2.73)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.74, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.75 to 1.24] — Effect of black tea adjusted for placebo

12. Other Pre Specified Outcome: Endothelium Independent Dilation, Chronic, Black Tea
Description: as for outcome 1
Time Frame: From before consumption on day 1 to before consumption day 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 9.55 (3.81) | 9.67 (3.37)
  Day 8, before consumption of test product | 9.86 (4.58) | 10.51 (4.16)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.41, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-2.12 to 0.88] — Effect of black tea adjusted for placebo

13. Other Pre Specified Outcome: Endothelium-Independent Dilation, Acute, Black Tea
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 1
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Arm/Group | Black Tea Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 9.55 (3.81) | 9.67 (3.37)
  Day 1, 2 hours post consumption of test product | 8.48 (3.66) | 8.28 (3.16)
Statistical Analysis 1: Comparison: Black Tea Beverage vs Placebo Beverage; Subject as random factor, baseline same period and mean baseline in both periods as covariates, and treatment, operator, and period as fixed effects; Test type: Superiority or Other; p = 0.74, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.11 to 1.54] — Effect of black tea adjusted for placebo

14. Other Pre Specified Outcome: Endothelium Independent Dilation, Acute-upon-chronic, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 8
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Groups:
- Postive Control Beverage: Participant when they received the positive control
Arm/Group | Postive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 10.05 (4.08) | 9.67 (3.37)
  Day 8, 2 hours post consumption of test product | 8.96 (3.69) | 9.28 (2.73)
Statistical Analysis 1: Comparison: Postive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.66, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.84 to 1.17] — Effect of positive control adjusted for placebo

15. Other Pre Specified Outcome: Endothelium Independent Dilation, Chronic, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to before consumption day 8
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 10.05 (4.08) | 9.67 (3.37)
  Day 8, before consumption of test product | 9.41 (3.98) | 10.51 (4.16)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-2.70 to 0.30] — Effect of positive control adjusted for placebo

16. Other Pre Specified Outcome: Endothelium Independent Dilation, Acute, Positive Control
Description: as for outcome 1
Time Frame: From before consumption on day 1 to 2 hours post consumption on day 1
Measure: Mean (Standard Deviation); unit: percentage of vascular dilation
Arm/Group | Positive Control Beverage | Placebo Beverage
Number analyzed (Participants) | 30 | 30
percentage of vascular dilation
  Day 1, before consumption of test product | 10.05 (4.08) | 9.67 (3.37)
  Day 1, 2 hours post consumption of test product | 8.74 (2.95) | 8.28 (3.16)
Statistical Analysis 1: Comparison: Positive Control Beverage vs Placebo Beverage; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.93 to 1.73] — Effect of positive control adjusted for placebo

ADVERSE EVENTS:
Time Frame: Three periods of one week intervention
Groups:
- Positive Control: Spray dried aqueous extract of a batch of tea extract that has shown to improve Flow Mediated Dilation previously
Arm/Group | Black Tea Extract | Positive Control | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 1/30 | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Black Tea Extract (N=30) | Positive Control (N=30) | Placebo (N=30)
Pyrexia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syncope (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No